CLINICAL TRIAL: NCT02209844
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses (2.5 mg to 1200 mg) of BI 44847 as Powder in the Bottle Reconstituted With 0.2% Natrosol Solution Administered to Healthy Male Subjects. A Randomised, Placebo-controlled (Within Dose Groups) and Double-blinded Trial
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses of BI 44847 Powder in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1224.1
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (2):
- BI 44847 powder (Experimental): single rising dose reconstituted with natrosol solution
  Interventions: Drug: BI 44847
- Placebo (Placebo Comparator): reconstituted with natrosol solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 44847
  Arms: BI 44847 powder
Drug: Placebo
  Arms: Placebo

SUMMARY:
To investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of BI 44847

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (BP, HR), 12-lead ECG, clinical laboratory tests
2. Age ≥ 18 and Age ≤ 50 years
3. BMI ≥ 18.5 and BMI ≤ 29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination (including BP, pulse rate and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
8. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
10. Participation in another trial with an investigational drug within two months prior to administration or during the trial
11. Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
12. Inability to refrain from smoking on trial days
13. Alcohol abuse (more than 60 g/day)
14. Drug abuse
15. Blood donation (more than 100 mL) within four weeks prior to administration or during the trial
16. Excessive physical activities (within one week prior to administration or during the trial)
17. Any laboratory value outside the reference range that is of clinical relevance
18. Inability to comply with dietary regimen of study centre
19. Any ECG value outside of the reference range and of clinical relevance including, but not limited to QRS interval > 120 ms. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval > 450 ms or QT> 500 ms).
20. A history of additional risk factors for Torsade des Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
21. The use of concomitant medications that prolong the QT/QTc interval
22. Elevated urinary glucose levels at screening (> 15 mg/dl)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2006-08; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to day 12
Number of patients with clinically significant findings in vital signs (blood pressure, pulse rate) | up to day 12
Number of patients with clinically significant findings in ECG | up to day 12
Number of patients with clinically significant laboratory findings | up to day 12
Assessment of tolerability by the investigator on a 4-point scale | up to day 12

SECONDARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | up to 96 hours after drug administration
tmax (time from dosing to maximum concentration) | up to 96 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 96 hours after drug administration
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | up to 96 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 96 hours after drug administration
λz (terminal rate constant in plasma) | up to 96 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 96 hours after drug administration
MRTpo (mean residence time of the analyte in the body after oral administration) | up to 96 hours after drug administration
CL/F (total clearance of the analyte in the plasma after extravascular administration) | up to 96 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 96 hours after drug administration
Aet1-t2 (amount of analyte that is eliminated in urine from the time point t1 to time point t2) | up to 72 hours after drug administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | up to 72 hours after drug administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 72 hours after drug administration
Area under the plasma glucose concentration time curve | up to 96 hours after drug administration
Total amount of glucose excreted in urine | up to 72 hours after drug administration
Maximum glucose concentration in plasma | up to 96 hours after drug administration
Maximum glucose concentration in urine | up to 72 hours after drug administration